CLINICAL TRIAL: NCT01189721
Title: Effect of Propofol on Remifentanil-induced Postoperative Hyperalgesia in Patients Undergoing Thyroid Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Gang nam Severance Hospital, Anesthesia and Pain Research Institute, Anesthesia and Pain Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2010-0102
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Hyperalgesia
Keywords: remifentanil; hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- sevoflurane (Active Comparator): Remifentanil will be infused intraoperatively at 0.2 ㎍/㎏/min. patients who are in this group will be infused propofol intraoperatively.
  Interventions: Drug: propofol, sevoflurane
- propofol (Experimental): Remifentanil will be infused intraoperatively at 0.2 ㎍/㎏/min. patients included this group will be inhaled sevoflurane intraoperatively.
  Interventions: Drug: propofol, sevoflurane

INTERVENTIONS:
Drug: propofol, sevoflurane — Remifentanil will be infused intraoperatively at 0.2 ㎍/㎏/min (group1 and 2) group 1 (Active Comparator, sevoflurane)will be infused propofol intraoperatively.
  group 2(Experimental, propofol) will be inhaled sevoflurane intraoperatively.

SUMMARY:
The investigators hypothesize that propofol infusion during surgery can affect the remifentanil hyperalgesia compared to sevoflurane inhalation.The outcome will be measured by a verbal numerical rating score (VNRS) and mechanical punctuating pain by electronic von frey filament.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thyroidectomy
* Age 20-65
* American Society of Anesthesiologists physical status classification I or II

Exclusion Criteria:

* History of chronic pain, Regular use of analgesic, antiepileptic or antidepressive drugs
* History of drug & alcohol abuse
* Psychiatric disorder
* Use of opioids within 24hrs
* Renal disease with decreased glomerular filtrate ratio
* Neuromuscular disease, Severe cardiac disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Tactile pain thresholds adjacent to the surgical wound assessed by von Frey hair before the induction and at postoperative 24 & 48 hrs | postoperative 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: yuen hee shim, MD, Study Chair — Gangnam severance hospital, Yonsei university, Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Reseach Institute
Locations (1):
- Gang Nam Severance Hospital, Yonsei University, Anesthesia and Pain Medicine Department,, Seoul, South Korea